CLINICAL TRIAL: NCT01283802
Title: More Than 400 Hepatectomies Without Intraoperative Cholangiography: Prospective Validation of the Role of Ultrasound
Brief Title: Intraoperative Cholangio-Ultrasound in Resective Liver Surgery
Acronym: IOCUS
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: GUIDO TORZILLI MD, PHD, UNIVERSITY OF MILAN
Other Study IDs: IOCUS
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2010-06

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IOCUS
  Interventions: Procedure: INTRAOPERATIVE CHOLANGIO-ULTRASOUND

INTERVENTIONS:
Procedure: INTRAOPERATIVE CHOLANGIO-ULTRASOUND — Techniques are as follows:
  1. Direct ultrasound exploration without any contrast agents.
  2. IOCUS injection into the bile duct of a mixture of air and saline (2 parts water and 1 part air);
  3. IOCUS injection of an air bolus into the bile duct.

SUMMARY:
Liver surgery should be considered an echo-guided procedure to guarantee conservative but radical resections. The investigators describe a further application of intraoperative ultrasonography (IOUS) for studying the biliary tree during liver surgery with no need for formal cholangiography.

DETAILED DESCRIPTION:
Intraoperative ultrasonography (IOUS) in liver surgery is widely accepted as a fundamental tool for radical and safe hepatectomy [1]. New technical improvements of IOUS have been reported in recent years both for tumor characterization and staging [2] and for resection guidance [3-5]. However, intraoperative cholangiography (IOC) still represents the gold standard for studying the biliary tract anatomy as well as for guiding reconstruction in case of bile duct resection and, moreover, with the advent of living donation it is the standard reference for validating preoperative imaging [6]. Conversely, it could be affirmed that IOUS in this sense has no role, if not for guiding intraoperative dilated bile duct drainage [7]. Nevertheless, IOC has not negligible costs, it implies the use of x-ray, iodated contrast agents and is time consuming.

Herein is proposed a technique for bile duct exploration by means of intraoperative cholangio-ultrasound (IOCUS) validated on a consecutive series of patients undergoing liver resection.

1. Machi J, Oishi AJ, Furumoto NL, Oishi RH (2004). Intraoperative ultrasound. Surg Clin North Am, 84(4): 1085-111
2. Minagawa M, Makuuchi M, Takayama T, Ohtomo K (2001). Selection criteria for hepatectomy in patients with hepatocellular carcinoma and portal vein tumor thrombus. Ann Surg, 233(3): 379-84
3. Torzilli G, Del Fabbro D, Olivari N, Calliada F, Montorsi M, Makuuchi M (2004). Contrast-enhanced intraoperative ultrasonography during liver surgery. Br J Surg, 91(9): 1165-7
4. Torzilli G, Makuuchi M. Ultrasound-guided finger compression in liver subsegmentectomy for hepatocellular carcinoma (2004). Surg Endosc, 18(1):136-9
5. Torzilli G, Takayama T, Hui AM, Kubota K, Harihara Y, Makuuchi M (1999). A new technical aspect of ultrasound-guided liver surgery. Am J Surg, 178(4): 341-3
6. Lee VS, Krinsky GA, Nazzaro CA, Chang JS, Babb JS, Lin JC, Morgan GR, Teperman LW. Defining intrahepatic biliary anatomy in living liver transplant donor candidates at mangafodipir trisodium-enhanced MR cholangiography versus conventional T2-weighted MR cholangiography. Radiology, 2004; 233(3): 659-66
7. Torzilli G, Makuuchi M, Komatsu Y, Noie T, Abe H, Kobayashi T, Kubota K, Takayama T. US guided biliary drainage during hepatopancreatico-jejunostomy for diffuse bile duct carcinoma. Hepatogastroenterology. 1999; 46(26): 863-6.

ELIGIBILITY:
Inclusion Criteria:

Patients who need:

* clarification of the bile duct anatomy;
* disclosure of eventual intrahepatic bile duct dilation;
* verification of the patency of a sutured bile duct after tumor detachment from a glissonian sheath;
* check of the drainage of a bile duct stump on the liver cut surface prior to bilio-enteric anastomoses.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing resective liver surgery for hepatobiliary tumors
Sampling Method: Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2004-06; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
the technical feasibility | 90- days for postoperative morbidity and mortality

SECONDARY OUTCOMES:
Efficacy | 90-days for postoperative morbidity and mortality
  Efficacy in providing the proper information validated by postoperative outcome and in particular by the absence of an undrained portion of the liver after resection, biliary reconstruction or bilio-enteric anastomoses, and the absence of consistent bile leaks

CONTACTS AND LOCATIONS:
Overall Officials: GUIDO TORZILLI, MD, PhD, Principal Investigator — University of Milan
Locations (1):
- Istituto Clinico Humanitas, Irccs, Rozzano - Milano, Italy

REFERENCES:
- [Background] Torzilli G, Donadon M, Marconi M, Palmisano A, Del Fabbro D, Spinelli A, Botea F, Montorsi M. Hepatectomy for stage B and stage C hepatocellular carcinoma in the Barcelona Clinic Liver Cancer classification: results of a prospective analysis. Arch Surg. 2008 Nov;143(11):1082-90. doi: 10.1001/archsurg.143.11.1082. PMID 19015467
- [Background] Torzilli G, Procopio F, Botea F, Marconi M, Del Fabbro D, Donadon M, Palmisano A, Spinelli A, Montorsi M. One-stage ultrasonographically guided hepatectomy for multiple bilobar colorectal metastases: a feasible and effective alternative to the 2-stage approach. Surgery. 2009 Jul;146(1):60-71. doi: 10.1016/j.surg.2009.02.017. PMID 19541011
- [Background] Torzilli G, Donadon M, Marconi M, Botea F, Palmisano A, Del Fabbro D, Procopio F, Montorsi M. Systematic extended right posterior sectionectomy: a safe and effective alternative to right hepatectomy. Ann Surg. 2008 Apr;247(4):603-11. doi: 10.1097/SLA.0b013e31816387d7. PMID 18362622
- [Background] Torzilli G, Montorsi M, Donadon M, Palmisano A, Del Fabbro D, Gambetti A, Olivari N, Makuuchi M. "Radical but conservative" is the main goal for ultrasonography-guided liver resection: prospective validation of this approach. J Am Coll Surg. 2005 Oct;201(4):517-28. doi: 10.1016/j.jamcollsurg.2005.04.026. PMID 16183489
- [Background] Torzilli G, Makuuchi M, Komatsu Y, Noie T, Abe H, Kobayashi T, Kubota K, Takayama T. US guided biliary drainage during hepatopancreatico-jejunostomy for diffuse bile duct carcinoma. Hepatogastroenterology. 1999 Mar-Apr;46(26):863-6. PMID 10370628